CLINICAL TRIAL: NCT06120231
Title: Pulse-width Modulation During Pedicle Screw Stimulation
Brief Title: Pulse-Width Modulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Linton T. Evans, Dr. Linton Evans, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY02001964
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-03

CONDITIONS: Spinal Fusion; Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pedicle Screw Stimulation Arm (Experimental)
  Interventions: Diagnostic Test: Pulse width modulation

INTERVENTIONS:
Diagnostic Test: Pulse width modulation — Will be stimulating the pedicle screws utilizing three different pulse-width settings, 0.4 milliseconds, 0.2 milliseconds, and 0.05 milliseconds.

SUMMARY:
The overarching aim of this project is to modulate the pulse-width during stimulation of pedicle screws and record the response thresholds associated with each PWM setting. During this initial phase of the investigation, no further data will be collected.

DETAILED DESCRIPTION:
In vivo electrical stimulation of pedicle screws is a well-documented modality for evaluating potential breach of the pedicle wall. However, previous research has focused primarily on the stimulation threshold intensity required to elicit a neurophysiological response. Other stimulation parameters, such as pulse-width, remain uninvestigated. The goal is to obtain data on the pulse-width vs. CMAP relationship.

ELIGIBILITY:
Inclusion Criteria:

* A patient will be eligible for study participation once they have been booked for a surgery involving pedicle screw placement and intraoperative neuromonitoring.

Exclusion Criteria:

* The study excludes neonates, minors, pregnant women, prisoners and cognitively impaired patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
CMAP response under three different pulse-width settings | Within operating room upon completion of pedicle screw placement. 1 day
  Upon completion of the pedicle screw placements, each screw will be stimulated utilizing three different pulse-width settings, 0.4 milliseconds, 0.2 milliseconds, and 0.05 milliseconds. The stimulation intensity required to elicit a compound muscle action potential (CMAP) will be recorded for each pulse-width parameter. This is measured in microvolts (uV).

CONTACTS AND LOCATIONS:
Overall Officials: Linton Evans, Dr., Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Health, Lebanon, New Hampshire, United States